CLINICAL TRIAL: NCT02693002
Title: Heart Failure Prevention for Women: Preservation of Cardiac Function in the Peri-Menopausal Woman Through Hormone Therapy
Brief Title: Estrogen Diastolic Heart Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment goals not being met
Sponsor: Gretchen Wells (Other)
Responsible Party: Sponsor-Investigator, Gretchen Wells, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-0798-F6A
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Menopause
MeSH Terms: interventions — estradiol, norethindrone drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hormone replacement therapy (Active Comparator): Estradiol/norethindrone acetate 1mg/0.5 mg by mouth oral daily for 12 weeks
  Interventions: Drug: Estradiol/Norethindrone acetate
- Placebo (Placebo Comparator): Inert ingredients by mouth oral daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estradiol/Norethindrone acetate — Estradiol/Norethindrone acetate 1mg/0.5 mg
  Other Names: Activella
  Arms: Hormone replacement therapy
Drug: Placebo — inactive ingredient
  Arms: Placebo

SUMMARY:
Peri-menopausal women will be randomized to hormone replacement therapy or placebo for 12 weeks to determine if markers of systolic and diastolic function change by echocardiography as well as laboratory markers of heart failure, including b-type natriuretic peptide (BNP).

DETAILED DESCRIPTION:
This preliminary, feasibility study will randomize 28 peri-menopausal women to either hormone replacement therapy or placebo for 12 weeks. Prior to randomization, each participant will undergo echocardiography, measurements of activity using the Duke Activity Status Index, measurements of quality of life and laboratory data, including b-type natriuretic peptide (BNP) measurements. Following the intervention for 12 weeks, these measurements will all be repeated.

ELIGIBILITY:
Inclusion Criteria:

* 28 healthy recently postmenopausal women with last menstrual bleeding 12 months at study entry. Women with last menstrual bleeding within 12 months at study entry are those who are peri-menopausal and for whom the drug is FDA approved.

Exclusion Criteria:

* History of hysterectomy, oophorectomy or both
* History of heart disease including cardiac transplantation, heart failure, bypass surgery or percutaneous intervention, and valve disease defined as moderate or severe valve regurgitation or stenosis
* History of bone disease including non-traumatic vertebral fractures on radiography
* Uncontrolled chronic disease (including uncontrolled diabetes defined as a hemoglobin A1C >8, uncontrolled hypertension defined as a systolic blood pressure >160 mmHg, awaiting organ transplant)
* Previous or current cancer, excluding basal cell carcinoma
* Previous or current thromboembolic disease
* Previous intolerance of Hormone replacement therapy (HRT) or Oral contraception (OC)
* Current or previous use of HRT within the past 3 months
* Current or recent (<12 months) substance abuse, including tobacco use
* No drug interactions with HRT
* No racial or ethnic groups will be excluded

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen L Wells, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be provided to participants of the study.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hormone Replacement Therapy | Placebo
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hormone Replacement Therapy | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Diastolic Function Assessed by Echocardiography
Description: Change in diastolic function as assessed by echocardiography from baseline to 12 weeks
Time Frame: Baseline and 12 weeks
Population: Data was not analyzed for this study. The study was terminated as a result of poor enrollment (N=1, Hormone replacement 1; N=2, placebo). Presenting data for such a low number of participants would compromise participant confidentiality.
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Activity Level Assessed by Duke Activity Status Index (DASI)
Description: Change in activity level as assessed by Duke Activity Status Index. The DASI estimates functional capacity through a series of 12 questions related to daily activity. Questions are scored as zero for a "No" answer or awarded a fixed number of points ranging from 1.75-8 for a "Yes" answer. Scores for each question are added, with the maximum score being 58.2 indicating a fully functional individual. Data are presented as the change in Mean score +/- SEM for each group at baseline and 12 weeks.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quality of Life Score Assessed by Utian Quality of Life Scale (UQoLS)
Description: Change in quality of life score as assessed by Utian Quality of Life scale. The UQoLS measures quality of life in four subcategories: Occupational, health, emotional and sexual. Questions are scored on a scale of 1-5 were 1 indicates "Not true of me" and 5 indicates an answer of "mostly true". Scores to the responses are added and evaluated within each subcategory. Higher scores indicate a higher quality of life within each subcategory with a maximum of 35 points for "Occupational", 31 points for "Health", 28 points for "Emotional" and 15 points for "Sexual" for a total of 100 points indicating the highest quality of life score possible. Data will be presented as the change in quality of life Mean +/- SEM over time.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: B-type Natriuretic Peptide (BNP) Levels
Description: Change in B-type natriuretic peptide (BNP) levels will be measure. Participants will have blood drawn via venipuncture and B-type natriuretic peptide will be measured using a quantitative chemiluminescent immunoassay. Data will be presented as the change in B-type natriuretic peptide over time.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Arm/Group | Hormone Replacement Therapy | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Hormone Replacement Therapy | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hormone Replacement Therapy (N=2) | Placebo (N=2)
Vaginal Bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Patient was randomized on 7/6/16. She developed vaginal bleeding on 8/7/16. Vaginal bleeding ICFinformed consent form. The patient underwent evaluation by primary care provider, stopped drug, and was withdrawn from the study.

LIMITATIONS AND CAVEATS:
Due to limited enrollment, there were too few participants to draw statistically meaningful conclusions from collected data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No